CLINICAL TRIAL: NCT06838416
Title: Evaluation of the Effect of Finerenone on Renal Function in Patients With Type 2 Diabetes and Chronic Kidney Disease: A Prospective, Single-Arm, Multicenter Clinical Study
Brief Title: Evaluation of the Effect of Finerenone on Renal Function in Patients With Type 2 Diabetes and Chronic Kidney Disease
Acronym: KSD-01
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: LK2023094; 00000000202109300008 (Other Grant/Funding Number: Shanghai Lingli Health Management Co., Ltd.)
Record Dates: First submitted 2025-02-17; First posted 2025-02-20 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes Mellitus; Chronic Kidney Disease; Renal Function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — finerenone; Angiotensin Receptor Antagonists

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Finerenone Treatment Group: All enrolled participants will receive finerenone as an add-on to their existing stable treatment regimen. The dose of finerenone will be adjusted based on eGFR levels at enrollment (10 mg once daily if eGFR < 60 mL/min/1.73 m²; 20 mg once daily if eGFR ≥ 60 mL/min/1.73 m²).
  Interventions: Drug: Finerenone

INTERVENTIONS:
Drug: Finerenone — Treatment will continue for 48 weeks.
  Other Names: Angiotensin II Receptor Blockers

SUMMARY:
Research Objectives To evaluate the impact of finerenone on renal function, diabetic complications, and safety in patients with Type 2 diabetes and chronic kidney disease.

Study Design Type: Prospective, single-arm, multicenter clinical trial. Sample Size: 300 patients. Intervention: Finerenone added to existing treatment regimen (10-20 mg once daily, dose adjusted based on eGFR), for 48 weeks.

Data Collection Time Points: Baseline, 4 weeks, 12 weeks, 24 weeks, 36 weeks, and 48 weeks.

Primary Endpoint: Change in urine albumin-to-creatinine ratio (UACR). Secondary Endpoints: Changes in eGFR, 24-hour urine protein, serum uric acid, retinopathy markers, pulse wave velocity (PWV), ankle-brachial index (ABI), etc.

Safety Endpoints: Changes in serum potassium, sodium, and blood pressure.

DETAILED DESCRIPTION:
Project Title Evaluation of the Effect of Finerenone on Renal Function in Patients with Type 2 Diabetes and Chronic Kidney Disease: A Prospective, Single-Arm, Multicenter Clinical Study The Objective of the Study

Primary Objective:

Evaluate the effect of finerenone on renal function in patients with Type 2 diabetes and chronic kidney disease.

Secondary Objectives:

Assess the impact of finerenone on the progression of diabetic retinopathy, diabetic peripheral vascular disease, and diabetic neuropathy in patients with Type 2 diabetes and chronic kidney disease.

Safety Objective:

Evaluate the general safety of finerenone in patients with Type 2 diabetes and chronic kidney disease.

Study Design This study is a prospective, single-arm, multicenter clinical trial conducted in patients with Type 2 diabetes and chronic kidney disease. It aims to evaluate the efficacy and safety of finerenone over a 48-week follow-up period, with a total of 300 participants.

Total number of patients 300 participants The Selection of patients

Inclusion Criteria:

Diagnosed with Type 2 diabetes according to the 1999 WHO criteria; aged ≥18 years; UACR ≥30 mg/g and eGFR ≥30 ml/min/1.73 m² sustained for over 3 months, with stable ARB/ACEI treatment for ≥4 weeks prior to enrollment; willing to sign a written informed consent and comply with the study protocol.

Exclusion Criteria:

Chronic kidney disease diagnosed before Type 2 diabetes. Serum potassium >4.8 mmol/L. Ineffective blood pressure control at screening (systolic BP ≥160 mmHg and/or diastolic BP ≥100 mmHg, average of three measurements in the supine position).

HbA1c >9%. Acute urinary tract infection or conditions affecting urine tests. Primary or secondary adrenal insufficiency. Use of mineralocorticoid receptor antagonists. Use of medications with clear effects on urine protein and eGFR within 4 weeks (except kininogenase).

Use of strong CYP3A4 inhibitors (e.g., itraconazole, ketoconazole, ritonavir, nelfinavir, cobicistat, clarithromycin, telithromycin, nefazodone, carbamazepine).

ALT or AST >2.5 × ULN, total bilirubin (TBIL) >2 × ULN. Use of systemic glucocorticoids for more than 7 days within 12 weeks prior to screening, or use of systemic glucocorticoids (intravenous/oral or intra-articular) or need for systemic immunosuppressive treatment within the past 14 days.

Any organ system cancer within the past 5 years, whether treated or untreated. Known pregnancy (positive pregnancy test), breastfeeding, recent plans for conception, or not using adequate contraception.

Participation in other interventional clinical trials within 3 months prior to screening.

Any severe systemic disease or other factors deemed inappropriate for study participation by the investigator.

Intervention Plan / Observation Plan On top of the existing stable treatment regimen, add Finerenone 10-20 mg once daily (qd). If eGFR <60 mL/min/1.73 m² at enrollment, administer 10 mg qd; if eGFR ≥60 mL/min/1.73 m², administer 20 mg qd. Continue treatment for 48 weeks.

Datas will be collected at baseline, 4 weeks, 12 weeks, 24 weeks, 36 weeks, and 48 weeks.

Evaluation Indicators

Primary Endpoint:

Change in Urine Albumin-to-Creatinine Ratio (UACR).

Secondary Endpoints:

Change in 24-hour urine protein quantification. Change in eGFR before and after treatment. Change in blood uric acid levels before and after treatment. Change in the number and area of retinal microaneurysms/hemorrhages, hard exudates, and cotton wool spots.

Change in pulse wave velocity (PWV). Change in Ankle-Brachial Index (ABI). Changes in echocardiographic measurements. Electromyography (EMG) (optional).

Safety Endpoints:

Serum potassium Serum sodium Blood pressure Statistical analysis Statistical analysis will be performed using R language. For normally distributed continuous data, mean ± standard deviation will be used for statistical description. For non-normally distributed data, median (P25, P75) will be used for statistical description. The comparison of quantitative data such as UACR before and after treatment will employ independent samples t-tests. Multivariate regression analysis will be conducted to assess the influencing factors of each endpoint.

Study Duration From October 1, 2023, to December 31, 2026

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 diabetes according to the 1999 WHO criteria
* Aged ≥18 years
* UACR ≥30 mg/g and eGFR ≥30 ml/min/1.73 m² sustained for over 3 months
* Stable ARB/ACEI treatment for ≥4 weeks prior to enrollment
* Willing to sign a written informed consent and comply with the study protocol

Exclusion Criteria:

* Chronic kidney disease diagnosed before Type 2 diabetes
* Serum potassium >4.8 mmol/L
* Ineffective blood pressure control at screening (systolic BP ≥160 mmHg and/or diastolic BP ≥100 mmHg, average of three measurements in the supine position)
* HbA1c >9%
* Acute urinary tract infection or conditions affecting urine tests
* Primary or secondary adrenal insufficiency
* Use of mineralocorticoid receptor antagonists
* Use of medications with clear effects on urine protein and eGFR within 4 weeks (except kininogenase)
* Use of strong CYP3A4 inhibitors (e.g., itraconazole, ketoconazole, ritonavir, nelfinavir, cobicistat, clarithromycin, telithromycin, nefazodone, carbamazepine)
* ALT or AST >2.5 × ULN, total bilirubin (TBIL) >2 × ULN
* Use of systemic glucocorticoids for more than 7 days within 12 weeks prior to screening, or use of systemic glucocorticoids (intravenous/oral or intra - articular) or need for systemic immunosuppressive treatment within the past 14 days
* Any organ system cancer within the past 5 years, whether treated or untreated
* Known pregnancy (positive pregnancy test), breastfeeding, recent plans for conception, or not using adequate contraception
* Participation in other interventional clinical trials within 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to evaluate the effects of finerenone on renal function and diabetic complications in patients with Type 2 diabetes mellitus (T2DM) and chronic kidney disease (CKD). The study population consists of adult patients diagnosed with T2DM and CKD who meet specific inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Urine Albumin-to-Creatinine Ratio (UACR) | Baseline to Week 48
  The primary outcome measure is the change in Urine Albumin-to-Creatinine Ratio (UACR) from baseline to the end of the 48-week treatment period. UACR is a key indicator of renal function and will be assessed to evaluate the efficacy of finerenone in reducing proteinuria in patients with Type 2 diabetes and chronic kidney disease.

SECONDARY OUTCOMES:
Change in eGFR | Baseline to Week 48
  The change in estimated Glomerular Filtration Rate (eGFR) from baseline to the end of the 48-week treatment period. eGFR is a key marker of renal function and will be used to assess the impact of finerenone on kidney function in patients with Type 2 diabetes and chronic kidney disease.
Change in 24-Hour Urine Protein Quantification | Baseline to Week 48
  The change in 24-hour urine protein quantification from baseline to the end of the 48-week treatment period. This measure will provide additional insight into the effect of finerenone on proteinuria in patients with chronic kidney disease.
Change in Blood Uric Acid Levels | Baseline to Week 48
  The change in serum uric acid levels from baseline to the end of the 48-week treatment period. Elevated uric acid levels are associated with renal dysfunction, and this measure will help assess the broader metabolic effects of finerenone.
Change in Pulse Wave Velocity (PWV) | Baseline to Week 48
  The change in pulse wave velocity (PWV) from baseline to the end of the 48-week treatment period. PWV is a measure of arterial stiffness and will be used to assess the impact of finerenone on cardiovascular health.
Change in Ankle-Brachial Index (ABI) | Baseline to Week 48
  The change in Ankle-Brachial Index (ABI) from baseline to the end of the 48-week treatment period. ABI is a measure of peripheral arterial disease and will be used to assess the impact of finerenone on peripheral vascular health.
Changes in Echocardiographic Measurements Title: Changes in Echocardiographic Measurements | Baseline to Week 48
  Changes in echocardiographic parameters (e.g., left ventricular mass index, ejection fraction) from baseline to the end of the 48-week treatment period. These measures will provide insights into the cardiovascular effects of finerenone in patients with Type 2 diabetes and chronic kidney disease.

CONTACTS AND LOCATIONS:
Overall Officials: Xie Ying, Ph.D., Principal Investigator — Second Affiliated Hospital of Suzhou University
Locations (1):
- The Second Affiliated Hospital of Suzhou University, Suzhou, Jiangsu, China